CLINICAL TRIAL: NCT00986375
Title: Online Program Assisting Lifestyle Changes: Adopting and Maintaining Physical Activity and Fruit & Vegetable Consumption (Asterix 1.0 & Obelix 2.0)
Brief Title: Online Program Assisting Lifestyle Changes (Asterix 1.0 & Obelix 2.0)
Acronym: OPAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Freie Universität Berlin (Other)
Responsible Party: Sonia Lippke, Dr.; Assistant Professor (C1), Freie Universität Berlin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FU-10-4711-001; Asterix_1.0; Obelix_2.0
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2011-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Randomized Controlled Trial; evidence- and theory-based behavioral intervention; expert system; stages of change; motivational interviewing; tailoring; Self Care; Rehabilitation; Expert Systems; Behavior; Motivation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (IG) (Experimental): Patients in the IG will receive an interactive, computerized expert system which tailors treatment components to the individual needs of the patients
  Interventions: Behavioral: Intervention Group (IG)
- Active Control Group (ACG) (Active Comparator): Patients in the ACG will get an interactive computerized standard program
  Interventions: Behavioral: Active Control Group (ACG)

INTERVENTIONS:
Behavioral: Intervention Group (IG) — patients will receive an interactive, computerized expert system which tailors treatment components to the individual needs of the patients
  Arms: Intervention Group (IG)
Behavioral: Active Control Group (ACG) — Patients in the ACG will get an interactive computerized standard program
  Arms: Active Control Group (ACG)

SUMMARY:
The purpose of this study is to help Internet users to adopt and maintain a healthy lifestyle, it is imperative to increase self-management competencies to improve healthy eating and regular physical activity. Aim of this research project is to evaluate an evidence- and theory-based computerized expert system in comparison to a standard program. In addition, two different tailoring criteria are compared to each other with regard to the misclassification of study participants. Internet users will be treated psychologically and followed up over 12 weeks. The computerized expert system is expected to help users better than the standard program. Both interventions are hypothesized to improve self-management competencies over time.

DETAILED DESCRIPTION:
Two experimental studies are planned over a time period of 12 weeks. In the nutrition study, participants will randomly be allocated to either a waiting control group (WCG) receiving a tailored intervention after the last follow-up questionnaire, an active control group (ACG), receiving an interactive quiz on all areas of healthy nutrition or to one of two intervention groups (IGs). Intervention group 1 receives one of four computerized tailored interventions based on a standard recommendation on vegetable and fruit intake, intervention group 2 receives one of the same four tailored interventions based on another criterion.

In the physical activity study, study participants in the intervention group receive an interactive, computerized expert system (Intervention Group, IG). Individuals in the Active Control Group (ACG) get a standard program, which does not tailor treatment components to the individual needs of the patients. Internet users (N = 1000) will be recruited in in the internet via press releases, personal invitations and advertised likes at well known web-sites. Study participants will be followed up over three measurement points: One to eight weeks after T1, T2 will take place. Four to 12 weeks after T1 the T3 measurement will be conducted.

The hypotheses are: Both the IG and the ACG are expected to have a higher motivation, to adopt a healthy lifestyle, to perform more health behavior and to be less likely to relapse into previous unhealthy routines at T2 and T3 than at T1. Also, IG and ACG will be healthier as well as they will report more quality of life and rehabilitation satisfaction at T2 and T3 than at T1. In comparison to ACG, the IG is hypothesized to be more effective than the ACG regarding motivation, behavior and social-cognitive predictors of behavior. Moreover, the interventions (ACG and IG) are supposed to be equally effective for different age and sex groups, obese and non-obese individuals. In the nutrition study, the IG2 will report higher on all outcome measures than IG1.

After successful evaluation and some adoptions the intervention will be implemented as a self-help program in all eligible Internet users in the Internet.

ELIGIBILITY:
Inclusion Criteria:

* to be capable of exercising on their own at a minimum level and/or to consume fruits and vegetables
* able to fill out a questionnaire (no illiteracy)
* adequate German language ability

Exclusion Criteria:

* no internet access
* no computer with keyboard

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
physical activity fruit & vegetable consumption | 12 weeks

SECONDARY OUTCOMES:
subjective health & well-being | 12 weeks
motivation/volition | 12 weeks
social-cognitive predictors of behavior (self-efficacy, action control etc.) | 12 weeks
intervention engagement | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Schwarzer, PhD, Study Chair — Freie Universitaet Berlin
Locations (1):
- Freie Universitaet Berlin, Berlin, State of Berlin, Germany